CLINICAL TRIAL: NCT00109941
Title: Treatment of Advanced Pancreatic Cancer With Opioid Growth Factor (OGF): Phase II
Brief Title: Opioid Growth Factor in Treating Patients With Advanced Pancreatic Cancer That Cannot Be Removed By Surgery
Acronym: OGF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000425404; FD-R-0002391 (Other Grant/Funding Number: FDA OOPD Grant FD-R-0002391); M01RR010732 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2013-03

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Enkephalin, Methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metenkephalin, OGF-opioid growth factor (Experimental): DRUG All subjects treated with met-enkephalin (also called OGF) 250 ug/kg iv weekly over 45 minutes
  Interventions: Biological: opioid growth factor; Biological: metenkephalin, OGF-opioid growth factor

INTERVENTIONS:
Biological: opioid growth factor — OGF was administered in saline at 250 ug/kg intravenously over 45 minutes
  Other Names: Opioid growth factor or OGF is a 5 amino acid peptide
Biological: metenkephalin, OGF-opioid growth factor — OGF given in saline iv 250 ug/kg weekly
  Other Names: opioid growth factor

SUMMARY:
RATIONALE: Opioid growth factor may stop the growth of pancreatic cancer by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well opioid growth factor works in treating patients with advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the growth inhibitory effects of opioid growth factor ([Met^5]-enkephalin) in patients with advanced unresectable pancreatic cancer.

Secondary

* Determine the pharmacokinetics of this drug in these patients.
* Determine the quality of life of patients treated with this drug.
* Determine the pain control, depression, and nutritional status of patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive opioid growth factor ([Met^5]-enkephalin) IV over 45 minutes once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 4 weeks during study treatment, and at the completion of study treatment.

Patients are followed weekly for survival.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of pancreatic cancer
* Advanced, unresectable disease
* Must have failed OR refused prior standard chemotherapy (e.g., gemcitabine or fluorouracil) for pancreatic cancer
* Measurable disease by radiography
* Age Over 18
* Performance status Karnofsky 50-100%
* Hematopoietic
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 3,500/mm^3
* Hemoglobin ≥ 8.5 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 4.0 mg/dL (stents allowed)
* PT or INR ≤ 2 seconds over control OR ≤ 1.8 (unless on warfarin) renal & metabolic
* BUN ≤ 30 mg/dL (hydrated)
* Creatinine ≤ 2.0 mg/dL
* Sodium ≥ 130 mmol/L
* Potassium ≥ 3.2 mmol/L
* Glucose 60-300 mg/dL
* Pulse 60-110 beats/minute
* Systolic blood pressure 90-170 mm Hg

Exclusion Criteria

* No primary CNS tumors or known brain metastases Cardiovascular
* - congestive heart failure
* symptoms of coronary artery disease
* cardiac arrhythmia
* poorly controlled hypertension
* myocardial infarction within the past year
* abnormal EKG
* asthma
* hronic obstructive pulmonary disease
* pregnant or nursing
* Fertile patients must use effective contraception
* serious infection requiring antibiotics within the past 2 weeks
* poorly controlled diabetes
* seizure disorders
* fever > 37.8° C
* other malignancy within the past 5 years
* concurrent chemotherapy
* concurrent oral steroids
* concurrent radiotherapy
* Surgery within 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Response (progressive disease, stable disease, partial response, complete response)
Tumor size
Quality of life
Depression
Opioid growth factor markers

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Smith, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Smith JP, Conter RL, Bingaman SI, Harvey HA, Mauger DT, Ahmad M, Demers LM, Stanley WB, McLaughlin PJ, Zagon IS. Treatment of advanced pancreatic cancer with opioid growth factor: phase I. Anticancer Drugs. 2004 Mar;15(3):203-9. doi: 10.1097/00001813-200403000-00003. PMID 15014352
- [Result] Smith JP, Bingaman SI, Mauger DT, Harvey HH, Demers LM, Zagon IS. Opioid growth factor improves clinical benefit and survival in patients with advanced pancreatic cancer. Open Access J Clin Trials. 2010 Mar 1;2010(2):37-48. doi: 10.2147/oajct.s8270. PMID 20890374